CLINICAL TRIAL: NCT06045026
Title: A Real-World Evidence Study Evaluating Oral Health Related Quality Of Life With Use Of A Stannous Fluoride Anti-Sensitivity Toothpaste For Dentin Hypersensitivity Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300058
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tin Fluorides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-sensitivity toothpaste (Other): Participants will use the anti-sensitivity toothpaste according to the instructions on the commercial pack and their normal oral healthcare habits for 24 weeks.
  Interventions: Other: Stannous fluoride

INTERVENTIONS:
Other: Stannous fluoride — Anti-sensitivity toothpaste containing 0.454% Stannous Fluoride

SUMMARY:
This study will evaluate the impact of long-term use of a desensitizing toothpaste containing 0.454 percent (%) stannous fluoride (SnF2) on oral health related quality of life (OHrQoL) in a population of self-reported dentin hypersensitivity (DH) sufferers. Data generated will provide real world information on the DH experience and DH management with a daily use anti-sensitivity treatment.

DETAILED DESCRIPTION:
This will be a decentralized, prospective, 24-week, monadic design, open label, study in a DH population. The study will evaluate changes in OHrQoL in participants with self-reported DH symptoms over 24 weeks of use of a DH treatment (anti-sensitivity toothpaste). OHrQoL will be measured using a validated questionnaire, the Dentin Hypersensitivity Experience Questionnaire (DHEQ-48), completed by study participants at Baseline, and Weeks 4, 8, 12, 16, 20, 24.

ELIGIBILITY:
Inclusion Criteria:

* Participant who has provided consent indicating they have been informed of all pertinent aspects of the study.
* All genders who, at the time of screening, are aged between 18 and 65 years (inclusive).
* Participant who is willing to complete all the assigned activities.
* Participant who is able to independently complete all the assigned activities on their smart devices.
* Participant who has tooth sensitivity (self-reported symptoms).

Exclusion Criteria:

* Participant whose sensitivity could be caused by other factors or clinical pathology than DH, as self-reported on the screening questionnaire, which include:

  1. Participant who has been/is on multiple prescription medications to treat severe acid reflux on a regular basis or has had surgery for acid reflux.
  2. Participant with full or partial denture(s).
  3. Participant who has undergone treatment for periodontal or gum disease within 6 months of screening or is currently undergoing treatment for periodontal or gum disease.
  4. Participant who has been informed by a Dental Health Care Professional (DHCP) that they have active periodontitis.
  5. Participant who has been informed by a DHCP that they have active caries.
  6. Participant with any chronic and/or severe painful health condition(s) which lead to regular use of pain relief medications (more than 3 days a week).
* Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ObvioHealth Virtual Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one decentralized center in the United States.
Pre-assignment Details: A total of 680 participants were screened, of which 536 participants were enrolled, and 460 participants completed the study. A total of 76 participants discontinued from the study.
Groups:
- Anti-sensitivity Toothpaste (Sensodyne Repair and Protect): Participants were instructed to brush their teeth (sensitive areas first) with anti-sensitivity toothpaste containing 0.454 percent (%) stannous fluoride (SnF2) for at least 1 minute twice daily (morning and evening, not more than 3 times a day) according to the directions on the commercial pack for up to 24 weeks.
Period: Overall Study
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Started | 536
Safety Population (Safety population included participants who completed at least 1 use of study product.) | 498
Modified Intent-to-treat (mITT) Population (mITT population included all participants who completed at least one use of study product and had at least 1 post-baseline derived Dentin Hypersensitivity Experience Questionnaire (DHEQ) total score.) | 491
Completed | 460
Not Completed | 76
Not completed — Lost to Follow-up | 60
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 3
Not completed — Enrollment closed | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included participants who completed at least 1 use of study product.
Groups:
- Anti-sensitivity Toothpaste (Sensodyne Repair and Protect): Participants were instructed to brush their teeth (sensitive areas first) with anti-sensitivity toothpaste containing 0.454% SnF2 for at least 1 minute twice daily (morning and evening, not more than 3 times a day) according to the directions on the commercial pack for up to 24 weeks.
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405
  Male | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58
  Not Hispanic or Latino | 437
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 265
  Black or African-American | 161
  Asian or Asian Indian | 38
  Mixed or Multiple Ethnic Groups | 24
  Other | 4
  American Indian or Alaska Native | 3
  Prefer not to answer | 3

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in DHEQ Total Score (Section 2, Question [Q]1-34) at Weeks 4, 8, 12, 16, 20 and 24
Description: The DHEQ is a condition-specific measure of oral-health related quality-of-life (OHrQoL) in relation to dentin hypersensitivity (DH). Section 2 of DHEQ included 34 questions grouped into 5 separate domains: Restrictions(Q1-4), Adaptation(Q5-16), Social Impact(Q17-21), Emotional Impact(Q22-29), and Identity(Q30-34). Participants scored each question using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score was derived from the sum of scores across all domains (Q1-34) and ranged from 34 to 238, where lower score indicated better quality of life in relation to DH. Change from Baseline was calculated by subtracting the Baseline score from the score at each indicated timepoint. A negative change from Baseline indicated improvement in OHrQoL.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: mITT population included all participants who completed at least one use of study product and had at least 1 post-baseline derived DHEQ total score. The Mixed Model with Repeated Measures (MMRM) included all participants in the mITT population in each analysis. Number analyzed represents the number of participants with non-missing data in the MMRM at the indicated timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -21.9 (1.52)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -35.4 (1.72)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -44.5 (1.94)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -51.6 (2.05)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -55.1 (2.12)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -62.0 (2.20)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

2. Primary Outcome: Adjusted Mean Change From Baseline in DHEQ Restrictions Domain (Section 2, Q1-4) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Restrictions domain of DHEQ evaluated 'the ways in which any sensations in teeth affected participants in their daily life'. It included 4 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 4 to 28. Lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting the Baseline score from the score at each indicated timepoint. A negative change from Baseline indicated improvement (less effect of sensations on participant's daily life).
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: mITT population. The MMRM included all participants in the mITT population in each analysis. Number analyzed represents the number of participants with non-missing data in the MMRM at the indicated timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -2.6 (0.20)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -4.7 (0.24)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -6.1 (0.27)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -7.2 (0.28)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -7.9 (0.29)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -8.5 (0.30)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

3. Primary Outcome: Adjusted Mean Change From Baseline in DHEQ Adaptation Domain (Section 2, Q5-16) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Adaptation domain of DHEQ evaluated 'the ways in which the sensations in teeth had forced participants to change things in their daily life'; 'things they did in their daily life to avoid experiencing the sensations in their teeth'. It included 12 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 12 to 84, where lower score indicated less effect of sensations on participant's daily life. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement (less effect of sensations on participant's daily life).
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -7.4 (0.58)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -12.6 (0.66)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -15.9 (0.73)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -18.6 (0.77)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -20.3 (0.79)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -22.9 (0.83)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

4. Primary Outcome: Adjusted Mean Change From Baseline in DHEQ Social Impact Domain (Section 2, Q17-21) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Social Impact domain of DHEQ evaluates 'the way the sensations affect participants when they are with other people or in certain situations.' It included 5 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 5 to 35, where lower score indicated less effect of sensations on participant's social life. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement (less effect of sensations on participant's social life).
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -2.9 (0.25)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -4.6 (0.29)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -5.7 (0.30)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -6.6 (0.31)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -7.2 (0.32)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -8.1 (0.33)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

5. Primary Outcome: Adjusted Mean Change From Baseline in DHEQ Emotional Impact Domain (Section 2, Q22-29) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Emotional Impact Domain of DHEQ evaluated 'the way the sensations in participant's teeth make them feel.' It included 8 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 8 to 56, where lower score indicated less impact of sensations on participant's emotions. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement in OHrQoL (less impact of sensations on participant's emotions).
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -6.2 (0.42)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -9.6 (0.47)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -11.6 (0.52)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -13.2 (0.54)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -13.6 (0.55)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -15.4 (0.58)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

6. Primary Outcome: Adjusted Mean Change From Baseline in DHEQ Identity Domain (Section 2, Q30-34) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Identity Domain of DHEQ evaluated 'what the sensations in participant's teeth mean for them.' It included 5 questions each scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranged from 5 to 35, where lower score indicated less impact of sensations on participant's identity. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement (less impact of sensations on participant's identity).
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -2.9 (0.29)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -3.9 (0.29)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -5.2 (0.33)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -5.9 (0.34)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -6.1 (0.35)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -7.1 (0.36)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

7. Secondary Outcome: Adjusted Mean Change From Baseline in Impact on Everyday Life (DHEQ Section 1, Q1-3) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: DHEQ Section 1 included 3 questions about participant's sensitive teeth and its impact on everyday life. Participants scored Q1 (how intense are the sensations?) on a scale of 1 (not at all intense) to 10 (worst imaginable); Q2 (how bothered are you by any sensations?) on a scale of 1 (not at all bothered) to 10 (extremely bothered); Q3 (how well can you tolerate sensations?) on a scale of 1 (can easily tolerate) to 10 (can't tolerate at all). The total score for each question ranged from 1 to 10; where lower scores indicated less intense, less bothersome and tolerable sensations. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement in intensity, botheration and tolerability of sensations.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Q1 (How intense are the sensations?): Change from Baseline at Week 4: number analyzed (Participants) | 488
  Q1 (How intense are the sensations?): Change from Baseline at Week 4 | -1.3 (0.07)
  Q1 (How intense are the sensations?): Change from Baseline at Week 8: number analyzed (Participants) | 483
  Q1 (How intense are the sensations?): Change from Baseline at Week 8 | -1.9 (0.07)
  Q1 (How intense are the sensations?): Change from Baseline at Week 12: number analyzed (Participants) | 474
  Q1 (How intense are the sensations?): Change from Baseline at Week 12 | -2.2 (0.07)
  Q1 (How intense are the sensations?): Change from Baseline at Week 16: number analyzed (Participants) | 471
  Q1 (How intense are the sensations?): Change from Baseline at Week 16 | -2.4 (0.08)
  Q1 (How intense are the sensations?): Change from Baseline at Week 20: number analyzed (Participants) | 453
  Q1 (How intense are the sensations?): Change from Baseline at Week 20 | -2.5 (0.08)
  Q1 (How intense are the sensations?): Change from Baseline at Week 24: number analyzed (Participants) | 460
  Q1 (How intense are the sensations?): Change from Baseline at Week 24 | -2.9 (0.09)
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 4: number analyzed (Participants) | 488
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 4 | -1.6 (0.08)
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 8: number analyzed (Participants) | 483
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 8 | -2.3 (0.09)
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 12: number analyzed (Participants) | 474
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 12 | -2.7 (0.09)
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 16: number analyzed (Participants) | 471
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 16 | -3.0 (0.09)
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 20: number analyzed (Participants) | 453
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 20 | -3.1 (0.09)
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 24: number analyzed (Participants) | 460
  Q2 (How bothered are you by any sensations?): Change from Baseline at Week 24 | -3.4 (0.09)
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 4: number analyzed (Participants) | 488
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 4 | -0.9 (0.08)
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 8: number analyzed (Participants) | 483
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 8 | -1.4 (0.08)
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 12: number analyzed (Participants) | 474
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 12 | -1.7 (0.09)
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 16: number analyzed (Participants) | 471
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 16 | -2.0 (0.09)
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 20: number analyzed (Participants) | 453
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 20 | -2.1 (0.09)
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 24: number analyzed (Participants) | 460
  Q3 (How well can you tolerate sensations?): Change from Baseline at Week 24 | -2.4 (0.09)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q1 (How intense are the sensations?): Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q1 (How intense are the sensations?): Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q1 (How intense are the sensations?): Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q1 (How intense are the sensations?): Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q1 (How intense are the sensations?): Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q1 (How intense are the sensations?): Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 7: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q2 (How bothered are you by any sensations?): Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 8: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q2 (How bothered are you by any sensations?): Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 9: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q2 (How bothered are you by any sensations?): Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 10: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q2 (How bothered are you by any sensations?): Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 11: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q2 (How bothered are you by any sensations?): Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 12: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q2 (How bothered are you by any sensations?): Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 13: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q3 (How well can you tolerate sensations?): Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 14: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q3 (How well can you tolerate sensations?): Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 15: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q3 (How well can you tolerate sensations?): Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 16: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q3 (How well can you tolerate sensations?): Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 17: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q3 (How well can you tolerate sensations?): Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 18: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Q3 (How well can you tolerate sensations?): Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

8. Secondary Outcome: Adjusted Mean Change From Baseline in Global Oral Health (DHEQ Section 2, Q35) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Global Oral Health was evaluated using a single question of DHEQ. Participants rated the overall health of their mouth, teeth, and gums using a 6-point scale ranging from 1 to 6 where 1=excellent, 2=very good, 3=good, 4=fair, 5=poor, and 6=very poor. Lower score indicated better oral health. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement in global oral health.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -0.1 (0.03)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -0.1 (0.03)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -0.2 (0.03)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -0.2 (0.04)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -0.3 (0.04)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -0.3 (0.04)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p = 0.0100, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

9. Secondary Outcome: Adjusted Mean Change From Baseline in Effect on Life Overall (DHEQ Section 2, Q36-39) Score at Weeks 4, 8, 12, 16, 20 and 24
Description: Effect on life was evaluated using 4 questions of DHEQ (Section 2, Q36-39) about how much the sensations in teeth affected participant's life overall. Participants scored each question on a 5-point scale ranging from 0 to 4 where 0=not at all, 1=a little, 2=somewhat; 3=quite a bit, and 4=very much. Thus, the total score ranged from 0 to 16, where lower score indicated less effect of sensations on participant's life overall. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement in overall quality of life (less effect of sensations on participant's life overall).
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 4: number analyzed (Participants) | 488
  Change from Baseline at Week 4 | -2.0 (0.14)
  Change from Baseline at Week 8: number analyzed (Participants) | 483
  Change from Baseline at Week 8 | -3.2 (0.15)
  Change from Baseline at Week 12: number analyzed (Participants) | 474
  Change from Baseline at Week 12 | -3.8 (0.17)
  Change from Baseline at Week 16: number analyzed (Participants) | 471
  Change from Baseline at Week 16 | -4.2 (0.17)
  Change from Baseline at Week 20: number analyzed (Participants) | 453
  Change from Baseline at Week 20 | -4.6 (0.17)
  Change from Baseline at Week 24: number analyzed (Participants) | 460
  Change from Baseline at Week 24 | -5.1 (0.17)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

10. Secondary Outcome: Percentage of Participants Who 'Agree' (Score 5-7) With Each Item (Statement) in the 5 DHEQ Domains (Section 2, Q1-34) at Baseline and Week 24
Description: The DHEQ is a condition-specific measure of OHrQoL in relation to DH. Section 2 of DHEQ included 34 questions grouped into 5 separate domains: Restrictions(Q1-4), Adaptation(Q5-16), Social Impact(Q17-21), Emotional Impact(Q22-29), and Identity(Q30-34). Participants scored each question using a 7-point scale ranging from 1(strongly disagree) to 7(strongly agree) where lower score indicated better quality of life in relation to DH. Scores 5 to 7 indicated agreement with the statement mentioned in the question, where 5=Agree a little, 6=Agree and 7=Strongly agree. Percentage of participants with scores 5 to 7 for each statement in the 5 DHEQ domains were reported.
Time Frame: Baseline (Week 0) and Week 24
Population: mITT population. Only those participants available at the indicated timepoints were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
percentage of participants
  Q1 (Restrictions): At Baseline | 95.5
  Q1 (Restrictions): At Week 24: number analyzed (Participants) | 460
  Q1 (Restrictions): At Week 24 | 48.0
  Q2 (Restrictions): At Baseline | 68.8
  Q2 (Restrictions): At Week 24: number analyzed (Participants) | 460
  Q2 (Restrictions): At Week 24 | 27.6
  Q3 (Restrictions): At Baseline | 85.7
  Q3 (Restrictions): At Week 24: number analyzed (Participants) | 460
  Q3 (Restrictions): At Week 24 | 36.7
  Q4 (Restrictions): At Baseline | 97.6
  Q4 (Restrictions): At Week 24: number analyzed (Participants) | 460
  Q4 (Restrictions): At Week 24 | 53.5
  Q5 (Adaptation): At Baseline | 96.3
  Q5 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q5 (Adaptation): At Week 24 | 46.1
  Q6 (Adaptation): At Baseline | 77.2
  Q6 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q6 (Adaptation): At Week 24 | 31.1
  Q7 (Adaptation): At Baseline | 87.2
  Q7 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q7 (Adaptation): At Week 24 | 40.4
  Q8 (Adaptation): At Baseline | 68.0
  Q8 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q8 (Adaptation): At Week 24 | 31.3
  Q9 (Adaptation): At Baseline | 69.5
  Q9 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q9 (Adaptation): At Week 24 | 35.9
  Q10 (Adaptation): At Baseline | 54.6
  Q10 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q10 (Adaptation): At Week 24 | 23.5
  Q11 (Adaptation): At Baseline | 89.0
  Q11 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q11 (Adaptation): At Week 24 | 41.3
  Q12 (Adaptation): At Baseline | 61.9
  Q12 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q12 (Adaptation): At Week 24 | 25.9
  Q13 (Adaptation): At Baseline | 92.5
  Q13 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q13 (Adaptation): At Week 24 | 48.7
  Q14 (Adaptation): At Baseline | 71.1
  Q14 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q14 (Adaptation): At Week 24 | 35.2
  Q15 (Adaptation): At Baseline | 79.8
  Q15 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q15 (Adaptation): At Week 24 | 38.0
  Q16 (Adaptation): At Baseline | 77.4
  Q16 (Adaptation): At Week 24: number analyzed (Participants) | 460
  Q16 (Adaptation): At Week 24 | 33.0
  Q17 (Social Impact): At Baseline | 73.3
  Q17 (Social Impact): At Week 24: number analyzed (Participants) | 460
  Q17 (Social Impact): At Week 24 | 30.9
  Q18 (Social Impact): At Baseline | 81.1
  Q18 (Social Impact): At Week 24: number analyzed (Participants) | 460
  Q18 (Social Impact): At Week 24 | 28.7
  Q19 (Social Impact): At Baseline | 58.0
  Q19 (Social Impact): At Week 24: number analyzed (Participants) | 460
  Q19 (Social Impact): At Week 24 | 23.9
  Q20 (Social Impact): At Baseline | 28.5
  Q20 (Social Impact): At Week 24: number analyzed (Participants) | 460
  Q20 (Social Impact): At Week 24 | 14.1
  Q21 (Social Impact): At Baseline | 75.4
  Q21 (Social Impact): At Week 24: number analyzed (Participants) | 460
  Q21 (Social Impact): At Week 24 | 44.8
  Q22 (Emotional Impact): At Baseline | 84.9
  Q22 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q22 (Emotional Impact): At Week 24 | 30.7
  Q23 (Emotional Impact): At Baseline | 91.0
  Q23 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q23 (Emotional Impact): At Week 24 | 43.3
  Q24 (Emotional Impact): At Baseline | 96.5
  Q24 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q24 (Emotional Impact): At Week 24 | 52.0
  Q25 (Emotional Impact): At Baseline | 66.2
  Q25 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q25 (Emotional Impact): At Week 24 | 33.7
  Q26 (Emotional Impact): At Baseline | 58.2
  Q26 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q26 (Emotional Impact): At Week 24 | 33.5
  Q27 (Emotional Impact): At Baseline | 98.2
  Q27 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q27 (Emotional Impact): At Week 24 | 55.9
  Q28 (Emotional Impact): At Baseline | 54.2
  Q28 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q28 (Emotional Impact): At Week 24 | 25.4
  Q29 (Emotional Impact): At Baseline | 81.5
  Q29 (Emotional Impact): At Week 24: number analyzed (Participants) | 460
  Q29 (Emotional Impact): At Week 24 | 35.4
  Q30 (Identity): At Baseline | 50.9
  Q30 (Identity): At Week 24: number analyzed (Participants) | 460
  Q30 (Identity): At Week 24 | 27.4
  Q31 (Identity): At Baseline | 60.9
  Q31 (Identity): At Week 24: number analyzed (Participants) | 460
  Q31 (Identity): At Week 24 | 32.4
  Q32 (Identity): At Baseline | 63.7
  Q32 (Identity): At Week 24: number analyzed (Participants) | 460
  Q32 (Identity): At Week 24 | 37.0
  Q33 (Identity): At Baseline | 63.7
  Q33 (Identity): At Week 24: number analyzed (Participants) | 460
  Q33 (Identity): At Week 24 | 32.8
  Q34 (Identity): At Baseline | 72.1
  Q34 (Identity): At Week 24: number analyzed (Participants) | 460
  Q34 (Identity): At Week 24 | 35.9

11. Secondary Outcome: Adjusted Mean Change From Baseline in Numeric Pain Rating Scale (NPRS) Score at Weeks 1, 2, 4, 8, 12, 16, 20 and 24
Description: NPRS was an 11-point segmented numeric version of a Visual Analogue Scale from which the participant selected a score from 0 to 10 that best reflected the intensity of their pain, where 0=no pain and 10=worst possible pain. Higher scores indicated of greater pain intensity. Change from Baseline was calculated by subtracting the Baseline score from score at each indicated timepoint. A negative change from Baseline indicated improvement (reduction in pain intensity).
Time Frame: Baseline (Week 0) and Weeks 1, 2, 4, 8, 12, 16, 20, 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
score on a scale
  Change from Baseline at Week 1: number analyzed (Participants) | 432
  Change from Baseline at Week 1 | -1.3 (0.09)
  Change from Baseline at Week 2: number analyzed (Participants) | 453
  Change from Baseline at Week 2 | -1.5 (0.09)
  Change from Baseline at Week 4: number analyzed (Participants) | 487
  Change from Baseline at Week 4 | -1.6 (0.09)
  Change from Baseline at Week 8: number analyzed (Participants) | 482
  Change from Baseline at Week 8 | -2.2 (0.09)
  Change from Baseline at Week 12: number analyzed (Participants) | 473
  Change from Baseline at Week 12 | -2.4 (0.10)
  Change from Baseline at Week 16: number analyzed (Participants) | 472
  Change from Baseline at Week 16 | -2.7 (0.10)
  Change from Baseline at Week 20: number analyzed (Participants) | 456
  Change from Baseline at Week 20 | -2.8 (0.10)
  Change from Baseline at Week 24: number analyzed (Participants) | 459
  Change from Baseline at Week 24 | -3.2 (0.10)
Statistical Analysis 1: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 1; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 2: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 2; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 3: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 4; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 4: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 8; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 5: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 12; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 6: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 16; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 7: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 20; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures
Statistical Analysis 8: Comparison: Anti-sensitivity Toothpaste (Sensodyne Repair and Protect); Change from Baseline at Week 24; Test type: Superiority; p < 0.0001, Mixed Model with Repeated Measures

12. Secondary Outcome: Satisfaction Numeric Rating Scale (NRS) Score at Week 24
Description: Participants were asked to rate their satisfaction with the DH treatment using NRS. NRS is an 11-point ordinal scale used to assess satisfaction with the overall management of the condition for which the participant sought help from treatment. The score ranged from 0 (completely dissatisfied) to 10 (completely satisfied), where higher scores indicated greater satisfaction with DH treatment.
Time Frame: Week 24
Population: mITT population. Here, overall number analyzed is defined as the number of participants with data available for analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 459
score on a scale | 7.8 (2.10)

13. Secondary Outcome: Number of Participants With Oral Hygiene Questionnaire (OHQ) Responses at Baseline
Description: Participants described their oral hygiene habits by completion of an OHQ. It included 9 questions: Q1:How frequently do you normally brush your teeth? Q2:Have you had a professional or self-applied tooth whitening treatment in the last 2 weeks? Q3:Have you had a professional tooth cleaning in the last 2 weeks? Q4:Have you ever been diagnosed with sensitive teeth by a dentist? Q5: When was the last time you visited a dentist/hygienist? Q6:Do you use a toothpaste designed specifically for sensitive teeth? Q7:What brand of toothpaste do you most frequently use? Q8:What type of toothbrush do you use? Q9:Can you tell me if you have any of the following: Cracked tooth/ teeth Chipped tooth/teeth, Cold sores, Grinding teeth, Gum swelling/inflammation, Receding gums, Painful/tender gums when brushing, Ulcers in the mouth, Stained/yellow teeth, Seeing blood when you spit when you brush your teeth, Bad breath, None of these. Number of Participants with OHQ Responses at Baseline were reported.
Time Frame: Baseline (Week 0)
Population: mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
Number analyzed (Participants) | 491
Participants
  Q1: How frequently do you normally brush your teeth? - 3 or more times a day | 47
  Q1: How frequently do you normally brush your teeth? - Twice a day | 394
  Q1: How frequently do you normally brush your teeth? - Once a day | 48
  Q1: How frequently do you normally brush your teeth? - Less Often | 2
  Q2: Have you had a professional or self-applied tooth whitening treatment in the last 2 weeks? -Yes | 2
  Q2: Have you had a professional or self-applied tooth whitening treatment in the last 2 weeks? - No | 489
  Q3: Have you had a professional tooth cleaning in the last 2 weeks? - Yes | 12
  Q3: Have you had a professional tooth cleaning in the last 2 weeks? - No | 479
  Q4: Have you ever been diagnosed with sensitive teeth by a dentist? - Yes | 183
  Q4: Have you ever been diagnosed with sensitive teeth by a dentist? - No | 308
  Q5: When was the last time you visited a dentist/hygienist? - Within 6 months | 256
  Q5: When was the last time you visited a dentist/hygienist? - Within the last year | 137
  Q5: When was the last time you visited a dentist/hygienist? - Within 2 years | 46
  Q5: When was the last time you visited a dentist/hygienist? - Between 2 and 3 years | 25
  Q5: When was the last time you visited a dentist/hygienist? - More than 3 years ago | 27
  Q6: Do you use a toothpaste designed specifically for sensitive teeth? - Yes | 91
  Q6: Do you use a toothpaste designed specifically for sensitive teeth? - No | 239
  Q6: Do you use a toothpaste designed specifically for sensitive teeth? - Sometimes | 149
  Q6: Do you use a toothpaste designed specifically for sensitive teeth? - Unknown | 12
  Q7: What brand of toothpaste do you most frequently use? - Act Toothpaste | 1
  Q7: What brand of toothpaste do you most frequently use? - Aquafresh Toothpaste | 3
  Q7: What brand of toothpaste do you most frequently use? - Arm & Hammer Toothpaste | 20
  Q7: What brand of toothpaste do you most frequently use? - Biotene Toothpaste | 1
  Q7: What brand of toothpaste do you most frequently use? - Burts Bees Toothpaste | 6
  Q7: What brand of toothpaste do you most frequently use? - Colgate Toothpaste | 168
  Q7: What brand of toothpaste do you most frequently use? - Crest Toothpaste | 157
  Q7: What brand of toothpaste do you most frequently use? - Hello Toothpaste | 9
  Q7: What brand of toothpaste do you most frequently use? - Jason Toothpaste | 2
  Q7: What brand of toothpaste do you most frequently use? - Orajel Toothpaste | 3
  Q7: What brand of toothpaste do you most frequently use? - Other Brand Toothpaste | 18
  Q7: What brand of toothpaste do you most frequently use? - Parodontax Toothpaste | 9
  Q7: What brand of toothpaste do you most frequently use? - Private Label Toothpaste | 6
  Q7: What brand of toothpaste do you most frequently use? - Rembrandt Toothpaste | 1
  Q7: What brand of toothpaste do you most frequently use? - Sensodyne Pronamel Toothpaste | 33
  Q7: What brand of toothpaste do you most frequently use? - Sensodyne Toothpaste | 38
  Q7: What brand of toothpaste do you most frequently use? - Therabreath Toothpaste | 2
  Q7: What brand of toothpaste do you most frequently use? - Toms Of Maine Toothpaste | 14
  Q8: What type of toothbrush do you use? - Manual toothbrush | 255
  Q8: What type of toothbrush do you use? - Power toothbrush | 137
  Q8: What type of toothbrush do you use? - Both - manual and power brushes | 99
  Q9: Can you tell me if you have any of the following? - Bad breath | 41
  Q9: Can you tell me if you have any of the following? - Chipped tooth or teeth | 51
  Q9: Can you tell me if you have any of the following? - Cold sores | 5
  Q9: Can you tell me if you have any of the following? - Cracked tooth or teeth | 19
  Q9: Can you tell me if you have any of the following? - Grinding teeth | 65
  Q9: Can you tell me if you have any of the following? - Gum swelling or inflammation | 23
  Q9: Can you tell me if you have any of the following? - None of these | 257
  Q9: Can you tell me if you have any of the following? - Painful/tender gums when brushing | 70
  Q9: Can you tell me if you have any of the following? - Receding gums | 41
  Q9: Can you tell me if you have any of the following? - Seeing blood when you spit/brush your teeth | 61
  Q9: Can you tell me if you have any of the following? - Stained/yellow teeth | 95
  Q9: Can you tell me if you have any of the following? - Ulcers in the mouth | 3

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) up to Week 24 (up to approximately 168 days)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a study participant, temporally associated with the use of a study product, whether or not considered related to the study product. A Serious AE (SAE) was a particular category of an AE where the adverse outcome was serious. All-Cause Mortality included all enrolled participants. Serious and Other AEs: Safety population included all participants who completed at least 1 use of study product.
Arm/Group | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect)
All-Cause Mortality (participants affected / at risk) | 0/536
Serious Adverse Events (participants affected / at risk) | 1/498
Other Adverse Events (participants affected / at risk) | 42/498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect) (N=498)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-sensitivity Toothpaste (Sensodyne Repair and Protect) (N=498)
Covid-19 (Infections and infestations) | 6
Upper Respiratory Tract Infection (Infections and infestations) | 4
Gingivitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Respiratory Tract Infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lyme Disease (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 1
Aphthous Ulcer (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 2
Dental Caries (Gastrointestinal disorders) | 1
Hyperaesthesia Teeth (Gastrointestinal disorders) | 1
Tooth Extraction (Surgical and medical procedures) | 2
Salpingectomy (Surgical and medical procedures) | 1
Wisdom Teeth Removal (Surgical and medical procedures) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Dandruff (Skin and subcutaneous tissue disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal Cyst (Renal and urinary disorders) | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1
Progesterone Decreased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT06045026/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT06045026/SAP_001.pdf